CLINICAL TRIAL: NCT07080957
Title: Comparative Outcomes of Mesh-Based and Mesh-Free Laparoscopic Uterus-Preserving Pectopexy for Apical Prolapse: A Retrospective Cohort Study
Brief Title: Comparison of Mesh-Based and Mesh-Free Laparoscopic Pectopexy in Uterus-Preserving Surgery for Apical Prolapse
Acronym: PectoMesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Havva Betül Bacak (Other Government)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, Specialist in Obstetrics and Gynecology, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gopMeshBasedMeshFreepecto
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: Laparoscopic Pectopexy; Apical Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: This is a single-center, retrospective cohort study designed to compare two surgical techniques-mesh-based and mesh-free laparoscopic uterus-preserving pectopexy-in patients diagnosed with apical pelvic organ prolapse. Data were collected from medical records of patients operated between 2021 and 2024. Participants were divided into two groups based on the type of surgical procedure received. Outcomes including anatomical correction, sexual function, operative time, complications, and recurrence were assessed using standardized instruments such as the POP-Q system and the PISQ-12 questionnaire. No randomization or blinding was applied due to the retrospective nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesh-free laparoscopic uterus-preserving pectopexy (Active Comparator): Patients in this group underwent laparoscopic uterus-preserving pectopexy without the use of synthetic mesh. Instead, native tissue fixation techniques were employed to achieve apical support. The uterus was preserved in all cases. Follow-up was conducted at 6 weeks, 3 months, and 1 year to evaluate outcomes.
  Interventions: Procedure: Mesh-free laparoscopic uterus-preserving pectopexy
- Mesh-based laparoscopic uterus-preserving pectopexy (Active Comparator): Patients in this group underwent laparoscopic uterus-preserving pectopexy using synthetic mesh for apical support. The mesh was fixed bilaterally to the iliopectineal ligaments to restore apical support while preserving the uterus. Outcomes were assessed preoperatively and at 6 weeks, 3 months, and 1 year postoperatively.
  Interventions: Procedure: Mesh-based laparoscopic uterus-preserving pectopexy

INTERVENTIONS:
Procedure: Mesh-free laparoscopic uterus-preserving pectopexy — Laparoscopic pectopexy without synthetic mesh was performed by utilizing native tissue fixation techniques. The uterus was suspended to the iliopectineal ligaments using permanent sutures without mesh implantation. The procedure aimed to provide apical support and avoid mesh-related complications. Postoperative follow-up included assessments of anatomical correction, functional recovery, and patient satisfaction.
  Arms: Mesh-free laparoscopic uterus-preserving pectopexy
Procedure: Mesh-based laparoscopic uterus-preserving pectopexy — Laparoscopic pectopexy was performed using a synthetic mesh to provide apical support while preserving the uterus. The mesh was bilaterally fixed to the iliopectineal (Cooper's) ligaments, and the uterus was suspended in a tension-free manner. This technique is designed to restore pelvic anatomy and improve symptoms of prolapse. Patients were followed postoperatively to assess anatomical success, complications, and functional outcomes.
  Arms: Mesh-based laparoscopic uterus-preserving pectopexy

SUMMARY:
This retrospective cohort study compares anatomical and functional outcomes of mesh-based and mesh-free laparoscopic uterus-preserving pectopexy in women with apical pelvic organ prolapse. A total of 81 patients were included between 2021 and 2024 (mesh-based: 41, mesh-free: 40). Key outcomes assessed included operative time, blood loss, hospital stay, anatomical correction (POP-Q), sexual function (PISQ-12), and complications. Both techniques significantly improved prolapse and sexual function. Mesh-based pectopexy offered superior apical and posterior support, while mesh-free pectopexy was associated with longer vaginal length and longer operative time. Complication and recurrence rates were low and similar across groups. The findings suggest that both techniques are effective, and surgical approach should be tailored to patient preference and clinical context.

DETAILED DESCRIPTION:
This retrospective cohort study was conducted to compare the anatomical and functional outcomes of mesh-based and mesh-free laparoscopic uterus-preserving pectopexy in the treatment of apical pelvic organ prolapse (POP). POP is a common condition among women, particularly those over 50 years of age, characterized by the descent of pelvic organs into the vaginal canal. While mesh-based procedures are known to offer robust apical support, they are associated with long-term complications such as mesh erosion, infection, and chronic pelvic pain. In contrast, mesh-free techniques may offer a safer alternative, particularly for patients wishing to avoid synthetic implants.

A total of 81 patients who underwent laparoscopic pectopexy between 2021 and 2024 at a tertiary care institution were included. Patients were divided into two groups based on the use of mesh: 41 underwent mesh-based and 40 underwent mesh-free procedures. Preoperative and postoperative assessments were conducted using the POP-Q (Pelvic Organ Prolapse Quantification) system for anatomical staging and the PISQ-12 (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire) for evaluating sexual function. Operative time, estimated blood loss, length of hospital stay, postoperative complications, and recurrence rates were also analyzed. Follow-up evaluations were scheduled at 6 weeks, 3 months, and 1 year.

The study found that both techniques significantly improved anatomical support and sexual function. Mesh-based pectopexy provided better apical and posterior compartment support, while the mesh-free approach resulted in a longer vaginal length and was preferred by patients seeking to avoid mesh-related complications. Operative time was significantly longer in the mesh-free group. Complication and recurrence rates were low and comparable between groups.

This study contributes to the growing body of evidence supporting uterus-preserving surgical options in POP treatment and highlights the importance of individualized surgical planning based on patient needs, preferences, and clinical profiles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pelvic organ prolapse (POP) classified as stage 2 or higher according to the POP-Q (Pelvic Organ Prolapse Quantification) system
* Desire for uterus preservation and refusal of hysterectomy during surgery
* Eligible for surgical intervention and able to undergo general anesthesia
* Women aged 18 years and older with pelvic organ prolapse

Exclusion Criteria:

* History of hysterectomy
* Severe comorbidities (e.g., serious cardiovascular diseases, bleeding disorders, or other medical conditions that may interfere with surgical treatment)
* Active infections in the pelvic or urogenital region
* Advanced malignancies (e.g., cancer)
* Psychological or cognitive impairments preventing informed consent or compliance with postoperative follow-up

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Anatomical Success According to POP-Q System | 1 year postoperatively
  Anatomical success is defined as apical pelvic support at stage 0 or I according to the Pelvic Organ Prolapse Quantification (POP-Q) system. Specific points evaluated include C (cervix or vaginal cuff), D (posterior fornix if applicable), Ba, Bp, and TVL (total vaginal length). Success indicates restored apical support without need for additional surgical intervention or evidence of recurrence at 1-year follow-up.
Change in Sexual Function Based on PISQ-12 Score | Baseline to 1 year postoperatively
  Sexual function was evaluated using the validated Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Scores range from 0 to 48, with higher scores indicating better sexual function. The primary endpoint was the change in total PISQ-12 score from baseline (preoperative) to 1 year postoperative. Improvements were compared between the mesh-based and mesh-free pectopexy groups to assess functional recovery related to sexual health.

CONTACTS AND LOCATIONS:
Overall Officials: enes serhat coşkun, md, Study Chair — University of Health Sciences, Gaziosmanpaşa Training and Research Hospital
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No